CLINICAL TRIAL: NCT02547168
Title: Determining the True Incidence of Atrial Fibrillation Before and After Lung Resection
Acronym: Lung-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial futility
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SJHH_Lung_AF
Record Dates: First submitted 2015-09-01; First posted 2015-09-11 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer; Atrial Fibrillation; Stroke
Keywords: Atrial Fibrillation; Symptomatic Atrial Fibrillation; Asymptomatic Atrial Fibrillation; Lung Resection; Ambulatory Cardiac Monitor
MeSH Terms: conditions — Lung Neoplasms; Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- iRhythm ZIO XT patch group (Experimental): This is the only arm in the study and patients within it will have a small, pebble shaped device adhered to their chests. This is an ECG (electrocardiogram) monitor and will measure the incidence of atrial fibrillation. It will have to be worn for 14 days before and after the lung resection procedure
  Interventions: Device: iRhythm ZIO XT patch

INTERVENTIONS:
Device: iRhythm ZIO XT patch — The iRhythm ZIO XT patch is an ECG monitor that has to be worn by study participants. It will be used to track any incidence of atrial fibrillation.

SUMMARY:
Lung resections for pulmonary malignancies offer the best chance of survival for patients, but these procedures carry a significant burden of post-operative morbidity and mortality. Patients are particularly at high risk for post-operative atrial fibrillation (a condition involving irregular heart rhythm). Atrial fibrillation with symptoms can increase the risk of stroke - a blockage in a major blood vessel in the brain, which can potentially result in a disability or even death. The objective of this study is to establish the feasibility of using ambulatory heart rate monitoring to determine the total incidence of atrial fibrillation in the peri-operative period before and after anatomic lung resection for malignancies. The study will also investigate the correlation between atrial fibrillation and rates of stroke and other adverse events, as well as serve to identify the patients that are at a higher risk of developing atrial fibrillation.

DETAILED DESCRIPTION:
Novel literature suggests that atrial fibrillation that is asymptomatic may just be as problematic as atrial fibrillation that presents itself with symptoms. The objective of the study is to establish the feasibility of tracking the total incidence of atrial fibrillation in the peri-operative period, including both symptomatic and asymptomatic events, using an ambulatory heart monitor. Additionally, the study aims to estimate the overall incidence of peri- and post-operative atrial fibrillation. These will be accomplished through usage of iRhythm ZIO XT, a small pebble shaped device that will be adhered to the patient's chest for 14 days before and after surgery, to measure how often atrial fibrillation occurs.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age and competent to consent
* Patients must be diagnosed with resectable lung cancer or metastatic lung disease eligible to complete metastasectomy
* Patients must have one of: Male gender, age greater than 65, hypertension, obesity, and recent tobacco use within the past year
* Patients must be booked for pneumonectomy, lobectomy or anatomical segmentectomy resection.

Exclusion Criteria:

* Patients undergoing emergent lung resection
* Patients undergoing lung resection for non-oncologic indications (lung biopsy, bullectomy)
* Patients with an existing neurostimulator
* Patients with pre-existing cardiac disease, defined as:

  * Patients with atrioventricular blockage of any degree or sick sinus syndrome;
  * Patients with known previous atrial fibrillation or flutter lasting more than 1 month;
  * Patients with any persistent diagnosed preoperative arrhythmia
  * Patients with implanted external defibrillators or pacemakers
* Patients with known adhesive allergies
* Inability to comply with or understand ambulatory monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Monthly rate of patient accrual | Ongoing from date of study initiation through to sample size completion, estimated to be 12 months
  Proportion of patients who are determined to be eligible for study relative to the number of patients actually enrolled and consented for participation in the study. This will help to inform the willingness of patients to participate in this study
Patient adherence to monitoring device use-Wear time | 28 day time period around lung resection
  Patient adherence to the device attachment requirements as stated in the study protocol, defined as the device remaining in place for at least 90% of the expected 28 day patch period (14 days before surgery and 14 days after) to determine feasibility of the study protocol in clinical context and patient tolerability. This will be measured by the iRhythm ZIO XT patch output.
Patient adherence to monitoring device use-Logging of symptomatic events | 28 day time period around lung resection
  Patient adherence to the symptomatic atrial fibrillation event logging task as stated in the study protocol, defined as the successful manual triggering of the device by the patient to note at least 80% of symptomatic events over the expected 28 day patch period (14 days before surgery and 14 days after) to determine feasibility of the study protocol in clinical context and patient tolerability. This will be measured by the iRhythm ZIO XT patch output.
Number of patients who withdraw from study protocol | 28 day time period around lung resection
  Number of patients who choose to withdraw from the study, defined as those who fail to complete the 14-day baseline monitoring period before surgery, decline to wear the device post-operatively, or drop out partway through the 14-day post-operative monitoring period. This will be measured by ongoing discussion with the patient and will help to determine the feasibility of the study protocol in clinical context and patient tolerability.

SECONDARY OUTCOMES:
Baseline incidence of asymptomatic atrial fibrillation before lung resection | Measured from 2 weeks preceding lung resection up to the day of procedure
  Number of unknown/asymptomatic/occult atrial fibrillation in the high-risk malignant lung resection population before surgery so that we know whether any differences in the event rate after surgery are likely to be as a result of the surgery itself. This will be measured by having patients wear the iRhythm ZIO XT patch for the 2 weeks before surgery
The number of post-operative atrial fibrillation events | Measured from post-operative day 1 to 14 days following lung resection
  Number of symptomatic and asymptomatic atrial fibrillation cases that occurred within 14 days of lung resection surgery, automatically measured by the iRhythm ZIO patch device for 2 weeks from the day after surgery
The number of any post-operative recurrent atrial fibrillation events within 14 days of lung resection | Difference in event rates between the 14 day baseline period before surgery and the 14 day period after surgery
  To compare the difference in post-operative atrial fibrillation rates between those who experienced any atrial fibrillation pre- and intra-operatively (recurrent atrial fibrillation) with those who did not as measured by a comparison of the two 14 day readings assessed by the iRhythm ZIO XT patch device.
Total event rate for asymptomatic atrial fibrillation | Comparison of the two intervals of 14 days preceding and 14 days following lung resection
  Number of asymptomatic atrial fibrillation events during the 28 day monitoring period, adjudicated by cardiology consultation of the ZIO XT patch output
Rate of other non- atrial fibrillation arrhythmia | Measured from post-operative day 1 to 14 days following lung resection
  Number of non- atrial fibrillation arrhythmias during the 14-day post-discharge time interval following lung resection, adjudicated by cardiology consultation of the ZIO XT patch output
Impact of resection intensity (larger versus smaller resection size) on the development of any atrial fibrillation events | Measured from post-operative day 1 to 14 days following lung resection
  Measure whether there is a difference in the number of recurrent, asymptomatic and/or symptomatic atrial fibrillation events depending on the amount of lung tissue removed as part of the resection, measured as per review of surgical characteristics noted in patient records
Impact of use of minimally invasive surgery on the development of any atrial fibrillation events | Measured from post-operative day 1 to 14 days following lung resection
  Measure whether there is a difference in the number of recurrent, asymptomatic and/or symptomatic atrial fibrillation events depending on whether an open or a minimally invasive technique was used to complete resection, measured as per review of surgical characteristics noted in patient records
Measurement of the difference of 90 day mortality in event-free patients and those with atrial fibrillation | Interval from the date of surgery to up to 90 days after surgery
  Number of deaths within 90 days of surgery, comparing between event-free and peri-operative atrial fibrillation sub-cohorts as determined by patient chart review
Measurement of the difference of rates of stroke in event-free patients and those with atrial fibrillation | Interval from the date of surgery to up to 90 days after surgery
  Number of strokes in untreated patients in the 30 and 90 day follow up periods, comparing between event-free and peri-operative atrial fibrillation cohorts as measured by the validated Questionnaire for Verifying Stroke-Free Status (QVSFS)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Shargall, MD FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No